CLINICAL TRIAL: NCT01545180
Title: Observatory: Search for Prognostic Factors of Pulmonary Hypertension Post-capillary in Heart Failure.
Acronym: PH-HF
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Collaborators: CHRU Lille, Dr Nicolas LAMBLIN (Unknown)
Responsible Party: Principal Investigator, Thibaud Damy, Assistant Professor, French Cardiology Society
Other Study IDs: 11415
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Post-capillary Pulmonary Hypertension
Keywords: Observatory; Heart failure; Post-capillary pulmonary hypertension; HTPcap
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 3 tubes of 6 blood for analysis of biomarkers
  * 2 tubes of 6 mL blood for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HTPcap in IC: HTPcap active and passive in a population of stable patients with heart failure (left ventricular ejection fraction impaired or preserved) and / or valvular disease who received a left right heart catheterization as part of their care.

SUMMARY:
This study will better understand the post-capillary pulmonary hypertension in heart failure, to determine its prognostic role and to consider specific treatment of different forms of pulmonary hypertension in post-capillary pulmonary heart failure.

DETAILED DESCRIPTION:
Patients with heart failure (HF) frequently have a post-capillary pulmonary hypertension (HTPcap) which has two forms: passive and reactive.

The prognosis, prevalence and pathophysiological mechanisms of cell and tissue involved in the onset and reversibility of these two forms of HTPcap remain poorly understood.

The latest recommendations of the European Society of Cardiology and the European Respiratory Society identify two forms of HTPcap in the IC as a function of the extent of trans-pulmonary gradient (GTP) measured during right heart catheterization (GTP = mPAP-Pcap): passive (GTP £ 12mmHg) and reactive (GTP> 12mmHg).

In the latter form, the increase in pulmonary pressure would be disproportionate to the increase in left ventricular pressures.

This study will permit to identify hemodynamic prognostic markers of the the IC, and clinical, biological and hemodynamic determinants of the HTPcap in the IC.

This will help to identify a population that could benefit from specific treatment to referred pulmonary artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with heart failure (LVEF preserved or altered or valvular heart disease) defined by a history of heart failure or LVEF less than or equal to 50%.
* Patient with a right heart catheterization for medical reasons
* Medical treatment considered optimal: beta blockers, ACE inhibitors or angiotensin II receptor antagonists and/or aldosterone
* Stable Patient: No significant cardiac decompensation or change the dose of diuretics for 28 days.
* The patient has agreed and have signed consent.

Exclusion Criteria:

* Patient is younger than 18 years.
* Patient with unstable heart failure (cardiogenic shock, acute cardiac decompensation).
* Coronary heart disease for which there is a maximum revascularization
* Organic valvular which is scheduled for surgical correction of valvular abnormality (plasty or replacement).
* Patient dialysis.
* PAH original pre-capillary catheterization, defined by a Pcap ≤ 15 mmHg.
* Patient with triple installation of PM within 90 days.
* Patients who underwent revascularization within 90 days.
* Patients who underwent mechanical ventricular assistance.
* Patient with severe lung infection (CPT < 60% of predicted, FEV < 60% predicted) or pulmonary embolism or respiratory failure with a paO2 in ambient air below 60mmHg or oxygen therapy.
* Patient with severe heart rhythm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of consecutive patients recruted from cardiology departments for all participating centres. Participation in the study is offered to all French institutions (academic hospitals, general hospitals, army hospitals and private clinics) with cardiology units. A physician is responsible for study recruitment at each centre.
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Prognostic | 2 years
  Estimate the prognosis of different forms of HTPcap in heart failure (ejection fraction altered, stored or valvular heart disease)

SECONDARY OUTCOMES:
Prevalence | 3 years
  Define the prevalence of different forms of active or passive HTPcap
Phenotype | 3 years
  Define the phenotypic characteristics of patients with reactive or passive HTPcap in heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud DAMY, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Cleland JG, Swedberg K, Follath F, Komajda M, Cohen-Solal A, Aguilar JC, Dietz R, Gavazzi A, Hobbs R, Korewicki J, Madeira HC, Moiseyev VS, Preda I, van Gilst WH, Widimsky J, Freemantle N, Eastaugh J, Mason J; Study Group on Diagnosis of the Working Group on Heart Failure of the European Society of Cardiology. The EuroHeart Failure survey programme-- a survey on the quality of care among patients with heart failure in Europe. Part 1: patient characteristics and diagnosis. Eur Heart J. 2003 Mar;24(5):442-63. doi: 10.1016/s0195-668x(02)00823-0. PMID 12633546
- [Background] Lainscak M, Cleland JG, Lenzen MJ, Follath F, Komajda M, Swedberg K. International variations in the treatment and co-morbidity of left ventricular systolic dysfunction: data from the EuroHeart Failure Survey. Eur J Heart Fail. 2007 Mar;9(3):292-9. doi: 10.1016/j.ejheart.2006.07.007. Epub 2006 Oct 4. PMID 17023204
- [Background] Metra M, Ponikowski P, Dickstein K, McMurray JJ, Gavazzi A, Bergh CH, Fraser AG, Jaarsma T, Pitsis A, Mohacsi P, Bohm M, Anker S, Dargie H, Brutsaert D, Komajda M; Heart Failure Association of the European Society of Cardiology. Advanced chronic heart failure: A position statement from the Study Group on Advanced Heart Failure of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2007 Jun-Jul;9(6-7):684-94. doi: 10.1016/j.ejheart.2007.04.003. Epub 2007 May 3. PMID 17481947
- [Background] Ghio S, Gavazzi A, Campana C, Inserra C, Klersy C, Sebastiani R, Arbustini E, Recusani F, Tavazzi L. Independent and additive prognostic value of right ventricular systolic function and pulmonary artery pressure in patients with chronic heart failure. J Am Coll Cardiol. 2001 Jan;37(1):183-8. doi: 10.1016/s0735-1097(00)01102-5. PMID 11153735
- [Background] Kjaergaard J, Akkan D, Iversen KK, Kjoller E, Kober L, Torp-Pedersen C, Hassager C. Prognostic importance of pulmonary hypertension in patients with heart failure. Am J Cardiol. 2007 Apr 15;99(8):1146-50. doi: 10.1016/j.amjcard.2006.11.052. Epub 2007 Mar 8. PMID 17437745
- [Background] Damy T, Viallet C, Lairez O, Deswarte G, Paulino A, Maison P, Vermes E, Gueret P, Adnot S, Dubois-Rande JL, Hittinger L. Comparison of four right ventricular systolic echocardiographic parameters to predict adverse outcomes in chronic heart failure. Eur J Heart Fail. 2009 Sep;11(9):818-24. doi: 10.1093/eurjhf/hfp111. PMID 19696055
- [Background] Damy T, Goode KM, Kallvikbacka-Bennett A, Lewinter C, Hobkirk J, Nikitin NP, Dubois-Rande JL, Hittinger L, Clark AL, Cleland JG. Determinants and prognostic value of pulmonary arterial pressure in patients with chronic heart failure. Eur Heart J. 2010 Sep;31(18):2280-90. doi: 10.1093/eurheartj/ehq245. Epub 2010 Aug 5. PMID 20693169
- [Background] Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G; ESC Committee for Practice Guidelines (CPG). Guidelines for the diagnosis and treatment of pulmonary hypertension: the Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS), endorsed by the International Society of Heart and Lung Transplantation (ISHLT). Eur Heart J. 2009 Oct;30(20):2493-537. doi: 10.1093/eurheartj/ehp297. Epub 2009 Aug 27. No abstract available. PMID 19713419
- [Background] Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT); Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G. Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2009 Dec;34(6):1219-63. doi: 10.1183/09031936.00139009. Epub 2009 Sep 12. No abstract available. PMID 19749199
- [Background] Moraes DL, Colucci WS, Givertz MM. Secondary pulmonary hypertension in chronic heart failure: the role of the endothelium in pathophysiology and management. Circulation. 2000 Oct 3;102(14):1718-23. doi: 10.1161/01.cir.102.14.1718. PMID 11015353
- [Background] Gehlbach BK, Geppert E. The pulmonary manifestations of left heart failure. Chest. 2004 Feb;125(2):669-82. doi: 10.1378/chest.125.2.669. PMID 14769751
- [Background] Wharton J, Strange JW, Moller GM, Growcott EJ, Ren X, Franklyn AP, Phillips SC, Wilkins MR. Antiproliferative effects of phosphodiesterase type 5 inhibition in human pulmonary artery cells. Am J Respir Crit Care Med. 2005 Jul 1;172(1):105-13. doi: 10.1164/rccm.200411-1587OC. Epub 2005 Apr 7. PMID 15817798
- [Background] Nagendran J, Archer SL, Soliman D, Gurtu V, Moudgil R, Haromy A, St Aubin C, Webster L, Rebeyka IM, Ross DB, Light PE, Dyck JR, Michelakis ED. Phosphodiesterase type 5 is highly expressed in the hypertrophied human right ventricle, and acute inhibition of phosphodiesterase type 5 improves contractility. Circulation. 2007 Jul 17;116(3):238-48. doi: 10.1161/CIRCULATIONAHA.106.655266. Epub 2007 Jul 2. PMID 17606845
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984
- [Background] Lewis GD, Shah R, Shahzad K, Camuso JM, Pappagianopoulos PP, Hung J, Tawakol A, Gerszten RE, Systrom DM, Bloch KD, Semigran MJ. Sildenafil improves exercise capacity and quality of life in patients with systolic heart failure and secondary pulmonary hypertension. Circulation. 2007 Oct 2;116(14):1555-62. doi: 10.1161/CIRCULATIONAHA.107.716373. Epub 2007 Sep 4. PMID 17785618
- [Background] Lewis GD, Lachmann J, Camuso J, Lepore JJ, Shin J, Martinovic ME, Systrom DM, Bloch KD, Semigran MJ. Sildenafil improves exercise hemodynamics and oxygen uptake in patients with systolic heart failure. Circulation. 2007 Jan 2;115(1):59-66. doi: 10.1161/CIRCULATIONAHA.106.626226. Epub 2006 Dec 18. PMID 17179022
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur Heart J. 2008 Oct;29(19):2388-442. doi: 10.1093/eurheartj/ehn309. Epub 2008 Sep 17. No abstract available. PMID 18799522